CLINICAL TRIAL: NCT02338817
Title: Clinical Evaluation of a Non-Invasive Hypoglycemia Detector in a Glycogen Storage Disease Population
Status: Terminated | Type: Observational
Why Stopped: The device often failed to detect hypoglycemic episodes in glycogen storage disease patients and the rate of false positive alarms was high.
Sponsor: University of Florida (Other)
Collaborators: Diabetes Sentry (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB201400105
Record Dates: First submitted 2014-12-11; First posted 2015-01-14 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Glycogen Storage Disease
MeSH Terms: conditions — Glycogen Storage Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GSD 1: These will be subjects with GSD I. The Diabetes Sentry device will be monitored for alarms for possible hypoglycemic. A blood sample will be taken to confirm blood glucose levels, lactate, and ketone values.
  Interventions: Device: Diabetes Sentry
- GSD 0, III, VI, or IX: These will be subjects with GSD 0, III, VI, or IX. The Diabetes Sentry device will be monitored for alarms for possible hypoglycemic. A blood sample will be taken to confirm blood glucose levels, lactate, and ketone values.
  Interventions: Device: Diabetes Sentry

INTERVENTIONS:
Device: Diabetes Sentry — The Diabetes Sentry device will be monitored for alarms for possible hypoglycemic. A blood sample will be taken to confirm blood glucose levels, lactate, and ketone values.
  Other Names: non-invasive hypoglycemia detector

SUMMARY:
Glycogen storage disease (GSD) patients frequently experience periods of hypoglycemia, putting them at risk for several complications, such as hepatomegaly, adenomas, and cirrhosis. As of now, glycogen storage disease patients are limited to using finger stick glucose meters to monitor their glycemia at home. Diabetes Sentry, a non-invasive hypoglycemia detector designed like a watch, has been available for diabetic patients to non-invasively alert for hypoglycemia, but has never been tested in a GSD population. The investigators propose to test the accuracy of the Diabetes Sentry on patients with GSD types 0, I, III, VI, and IX, by measuring their metabolic markers every two hours, as well as whenever the device alerts for hypoglycemia. If accurate, it could be a useful tool for GSD patients in managing hypoglycemia, both clinically and at home.

DETAILED DESCRIPTION:
As a participant the following will take place:

The Diabetes Sentry device, which is non-invasive and is worn on the wrist will be used while an inpatient at the University of Florida Health & Shands Hospital. Participants will be monitored for the duration of the observational period on the unit, an expected average will be 24 hours. The device is designed to alarm during periods of perspiration and drops in body temperature. When this occurs, a blood draw will be taken to test for glucose, lactate, and ketone values at those times if there is not an already scheduled clinical care blood draw for normal clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed and clinically treated at the University of Florida with any of the glycogen storage diseases I, III, VI, IX, 0 will be asked to participate in this study.

Exclusion Criteria:

* Patients not clinically treated at the University of Florida.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed and clinically treated at the University of Florida with any of the glycogen storage diseases
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | At time of alarm (Average of 24 hours)
  glucose level at time of device alarm
Blood Lactate | At time of alarm (Average of 24 hours)
  lactate level at time of device alarm
Blood Ketones | At time of alarm (Average of 24 hours)
  ketone level at time of device alarm

CONTACTS AND LOCATIONS:
Overall Officials: David A Weinstein, MD, MMSc, Principal Investigator — Univeristy of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States